CLINICAL TRIAL: NCT03271853
Title: Thermalogical Analysis of a Cohort of Women and Men Undergoing Mammographic Analysis.
Status: Suspended | Type: Observational
Why Stopped: Trial temporarily halted to conduct additional device testing to verify cooling data. This temporary halt is NOT due to a potential risk to subject safety.
Sponsor: First Sense Medical, LLC (Other)
Collaborators: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Other Study IDs: SBS-001
Record Dates: First submitted 2017-07-24; First posted 2017-09-05 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Breast Neoplasm Female; Cancer, Breast; Thermography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- SBS II
  Interventions: Device: Sentinel BreastScan II

INTERVENTIONS:
Device: Sentinel BreastScan II — The SBS II will automate the recording of thermal data used in the Therma-Scan manual thermology protocol by utilizing a thermal camera sensitive to changes in breast temperature. The SBS II system uses a very sensitive thermography camera that detects and visually displays heat patterns that naturally emanate from the breast. SBS II captures this data digitally for subsequent analysis by Therma-Scan.

SUMMARY:
This study is designed to evaluate the Sentinel BreastScan II as well as the analysis of data by Therma-Scan.

DETAILED DESCRIPTION:
FirstSense Medical, LLC is a medical device company which has developed a breast cancer screening device, the Sentinel BreastScan II [SBS II]. This radiation free device is being developed to produce data which will be analyzed by Therma-Scan Reference Laboratory. Dr. Hoekstra, CEO of Therma-Scan, is the author of a published paper based on breast thermal data with a reported 95% sensitivity and 91% specificity. The SBS II examination will take approximately 7 minutes.

This study is designed to evaluate the Sentinel BreastScan II as well as the analysis of data by Therma-Scan. SBS II thermal breast data is an adjunctive aid to standard breast imaging. Currently, mammography is one of the standards of care in screening for visible signs of breast cancer. Breast thermology is the analysis of the heat signature data from an examined breast. All study costs will be incurred by the sponsor. Study subjects will incur no cost to participate. All scientific data revealed in this protocol will be used for the specific objectives of the study. The SBS II is a non-significant risk device. There is no contact with the subject during the entire procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, over the age of 18 years of age.
* Asymptomatic women or women who are being screened for breast abnormality.
* Women scheduled for a mammogram or women who have had a mammogram and are given 3 days to wait in between their mammogram and scheduled biopsy and FS/TS system.
* Not pregnant or breast feeding.
* Signed Informed consent.

Exclusion Criteria:

* Subject does not meet inclusion criteria, noted above.
* Use of 100 mg or more of niacin by tablet or niacin patch within the last 24 hours.
* Use of nitroglycerin within the last 24 hours.
* Subject experienced a fever of 102°F or higher within thirty-six (36) hours of the study.
* Subject must not have had a mammogram, breast ultrasound, or breast exam within the last 72 hours prior to the SBS II.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male or Female, over the age of 18 years.
Study Population: Study population consists of any patient undergoing standard mammographic examination and/or any additional imaging study predicated on the results of mammography.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-03 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Measure protocol accuracy | Through study completion, an average of 4 years.
  To measure the sensitivity and specificity of thermographic analysis based on the Marseilles analytic protocol [ Th 1 thru 5 ] to biopsy results predicated on standard breast imaging criteria [ BIRADS analytical protocol, B1 thru B5 ]. The resultant BIRADS score and biopsy pathological results will be compared to thermographic analysis [ Th1 thru 5 ] for each subject. 50 subjects undergoing both thermography and standard breast imaging leading to biopsy [ BIRADS 3 thru 5 ] will then be compared by measuring the results of each, BIRADS for standard breast imaging v the Marseilles Th system used in thermographic analysis, for concordance or discordance of findings as measured on final pathological analysis. This analysis will be performed for each subsequent 50 patient cohort undergoing standard mammographic/ultrasound breast imaging analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Elsamaloty, Principal Investigator — University of Toledo
Locations (1):
- Eleanor N. Dana Cancer Center, University of Toledo, Toledo, Ohio, United States

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03271853/Prot_000.pdf
  • Informed Consent Form (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT03271853/ICF_001.pdf